CLINICAL TRIAL: NCT06171555
Title: Efficacy of Connective Tissue Allograft Versus Steroid Injections in Treatment of Lateral Epicondylitis
Brief Title: Efficacy of CTM for Tennis ELbow
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Indiana Hand to Shoulder Center (Other)
Collaborators: CTM Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHTSC CTM Project HC22-1
Record Dates: First submitted 2023-11-30; First posted 2023-12-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-12

CONDITIONS: Tennis Elbow; Lateral Epicondylitis (Tennis Elbow); Lateral Elbow Tendinopathy
MeSH Terms: conditions — Tennis Elbow | interventions — Betamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Group 1 Control Group: standard corticosteroid injection: 1cc of celestone (6mg) diluted with 1 cc of 1% lidocaine and inject at the ECRB origin at area of maximal pain when palpated.
  Group 2 Test Group: CTM injection: 1cc of CTM Boost will be diluted with 1 cc of 1% lidocaine and injected at the ECRB origin at area of maximal pain when palpated. CTM Boost is a connective tissue matrix suspended in saline. (injection will need to be with a 23 gauge needle and 3 cc syringe)
  Randomization will be through a computerized random allocation assigned by the Research Coordinator on the day of consent.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care Steroid Injection (Active Comparator): Group 1 Control Group: standard corticosteroid injection: 1cc of celestone (6mg) diluted with 1 cc of 1% lidocaine and inject at the ECRB origin at area of maximal pain when palpated.
  Interventions: Drug: Celestone
- Test CTM Injection (Experimental): Group 2 Test Group: CTM injection: 1cc of CTM Boost will be diluted with 1 cc of 1% lidocaine and injected at the ECRB origin at area of maximal pain when palpated. CTM Boost is a connective tissue matrix suspended in saline. (injection will need to be with a 23 gauge needle and 3 cc syringe)
  Interventions: Device: CTM

INTERVENTIONS:
Device: CTM — decellularized particulate human placental connective-tissue matrix products, intended solely for homologous use to supplement or replace damaged or inadequate connective-tissue. These are structural tissue allografts processed according to the criteria contained in 21CFR 1271.10(a) for regulation solely under section 361 of the Public Health Service Act.
  Other Names: Connective Tissue Matrix
  Arms: Test CTM Injection
Drug: Celestone — standard of care
  Other Names: Corticosteroid
  Arms: Standard of Care Steroid Injection

SUMMARY:
In this study, the objective is to evaluate the effectiveness of a single application of human Connective Tissue Allograft (CTA) as a treatment of LET. CTM Biomedical markets and distributes decellularized particulate human placental connective-tissue matrix products, intended solely for homologous use to supplement or replace damaged or inadequate connective-tissue. These are structural tissue allografts processed according to the criteria contained in 21CFR 1271.10(a) for regulation solely under section 361 of the Public Health Service Act. Drug/Device Handling: If the research involves drugs or device, describe your plans to store, handle, and administer those drugs or devices so that they will be used only on subjects and be used only by authorized investigators.

DETAILED DESCRIPTION:
Lateral Elbow Tendinopathy (LET) is considered an overload injury of the extensor tendons of the forearm where they attach at the lateral epicondyle. LET is a common condition encountered both in primary care and specialty clinics. A population-based study reported an incidence of 3.4 (95% CI, 3.3-3.5) per 1000. The highest incidence was among individuals aged 40 to 49 years, with 7.8 per 1000 in male patients and 10.2 per 1000 in female patients. Work restrictions were reported in 16% of the patients, and 4% reported missing 1 to 12 weeks of work. The recurrence rate within 2 years was 8.5% and remained constant over time. The study data suggest that patients without resolution after 6 months of onset may have a prolonged disease course and may need surgical intervention. The patient demographic is typically active in the workforce and LET related absenteeism results in a substantial economic impact. Pain relief, timely return to work, and avoidance of surgical intervention are therefore important LET treatment goals. Patients suffering from LET are grouped into 2 entities: Group 1 experience symptoms in an acute (tendinitis) phase that is largely influenced by the local inflammation stemming from over-use activities. Group 2 developed tendon degeneration and/or bony responses due to a persistent, chronic (tendinosis) pathology. Histologic specimens from chronic cases confirm that tendinosis is not an acute inflammatory condition but rather a failure of the normal tendon repair mechanism associated with angio-fibroblastic degeneration. The cause of elbow tendinosis is most likely a combination of mechanical overloading and abnormal microvascular responses. Further research into the precise cause of tendinosis is, however, still needed. The chief complaint in both groups is elbow pain with or without activity. Numerous methods have been advocated for treating LET including rest, nonsteroidal anti-inflammatory medication, bracing, physical therapy, iontophoresis, extracorporeal shock wave therapy, and botulism toxin. Injections of corticosteroids or whole blood, and various types of surgical procedures have also been recommended. The utility of several of these treatments has recently come into question. For example, one recent report noted that there is no difference between using corticosteroid or local anesthetic when treating elbow tendinosis with an injection. A recent review of common growth factors suggested human CTA may be useful for tendon and ligament healing in vivo.

The primary study endpoint is based on the hypothesis that treatment of LET with a single application of CTA will provide a clinically meaningful improvement of the Patient-Related Tennis Elbow Evaluation (PRTEE) Pain Subscale Secondary endpoints include VAS pain and elbow range of motion. Secondary endpoints also include PROMIS scores of pain interference and depression. A single assessment numerical evaluation (SANE) of elbow function will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 or older
2. Patients presenting with symptomatic lateral epicondylitis for at least 6 weeks
3. Patients who have not had a meaningful symptomatic improvement after 6 weeks of physical therapy
4. Patients who can consent to be a part of this study
5. Patients who are able to return to the Indiana Hand to Shoulder Center or a satellite location for follow up time points

Exclusion Criteria:

1. Previous surgery to the lateral side of the elbow
2. Systemic inflammatory conditions (RA, psoriatic arthritis, lupus, etc)
3. Previous elbow injection within the last 6 months
4. History of recent elbow trauma
5. Patients actively involved in workman's compensation cases
6. Non-English Speaking Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Related Tennis Elbow Evaluation (PRTEE) Pain Subscale | 6 Months
  PROM

SECONDARY OUTCOMES:
VAS Pain | 6 Months
  pain
PROMIS Pain Interference | 6 Months
  PROM
PROMIS Depression | 6 Months
  PROM
Grip Strength | 6 Months
  grip strength taken with a calibrated jamar instrument
Range of Motion | 6 Months
  wrist range of motion measured with a goniometer with elbow both flexed and extended

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No